CLINICAL TRIAL: NCT05023512
Title: Together Researching Understanding, Solidarity, and Trust Around COVID - TRUST Study
Brief Title: Understanding Public Attitudes Towards the COVID-19 Vaccination
Acronym: CEAL
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: This study is not a clinical trial.
Sponsor: University of Massachusetts, Worcester (Other)
Collaborators: Boston University (Other); National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Kimberly Fisher, Associate Professor, University of Massachusetts, Worcester
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Prevention
Other Study IDs: H00023672; 1OT2HL156812-01 (NIH)
Record Dates: First submitted 2021-08-24; First posted 2021-08-26 (Actual); Last update posted 2022-06-06 (Actual); Status verified 2022-06

CONDITIONS: Covid19; Vaccination
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Message 1 (Experimental): Participants will be randomized to receive version #1 of 2 different versions of a message from the Massachusetts Department of Public Health regarding the COVID-19 vaccination.
  Interventions: Behavioral: Communication about the COVID-19 vaccination from the Massachusetts Department of Public Health
- Message 2 (Experimental): Participants will be randomized to receive version #2 of 2 different versions of a message from the Massachusetts Department of Public Health regarding the COVID-19 vaccination.
  Interventions: Behavioral: Communication about the COVID-19 vaccination from the Massachusetts Department of Public Health

INTERVENTIONS:
Behavioral: Communication about the COVID-19 vaccination from the Massachusetts Department of Public Health — Participants will be randomized to receive one of two different versions of messages from the Massachusetts Department of Public Health. The message that participants in each experimental group receive will vary slightly and systematically. Specific content and wording of these messages were developed to address and mitigate concerns about the Covid-19 vaccination.

SUMMARY:
The objective of this study is to better understand public attitudes towards coronavirus disease 2019 (COVID-19) vaccination. This understanding will inform the development of community engagement strategies to be used in future interventions and studies aimed at addressing factors that impact the disproportionate burden of COVID-19 in under-served and vulnerable communities.

DETAILED DESCRIPTION:
The severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2) has rapidly instigated a global pandemic. As of this writing, there are more than 33 million documented cases of infection in the United States (US). Furthermore, in the US, COVID-19 has disrupted the economy, overwhelmed the healthcare system, led to widespread school cancellations, and caused more than 595,000 deaths since March 2020.

The availability of three highly effective vaccines against COVID-19 within a year of the start of the pandemic is an extraordinary achievement and cause for great optimism. However, a significant proportion of adults in the U.S. have not accepted vaccination against COVID-19. Efforts are needed to identify effective messages and communication strategies to overcome COVID-19 vaccine hesitancy.

To address this need, the investigators plan to conduct two rapid surveys among Massachusetts residents, to assess attitudes towards COVID-19 vaccination.

ELIGIBILITY:
Inclusion Criteria:

* Massachusetts resident
* Adult (age 18 and over)
* English or Spanish speaking

Exclusion Criteria:

• Non-English or Spanish speaking

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2021-10-28 (Actual); Primary Completion 2022-07-15 (Estimated); Study Completion 2022-09-01 (Estimated)

PRIMARY OUTCOMES:
Intent to be vaccinated against Covid-19 among unvaccinated participants | Through survey completion, an average of 12 minutes
  The survey includes a question that assesses participants' willingness to be vaccinated against Covid-19 if they are unvaccinated. Responses include Yes, No, or Not Sure to being vaccinated against Covid-19.

CONTACTS AND LOCATIONS:
Overall Officials: Kimberly Fisher, MD, Principal Investigator — University of Massachusetts, Worcester

IPD SHARING:
Plan to Share IPD: No